CLINICAL TRIAL: NCT06098131
Title: Comparative Effects of the Neurodynamic Slider and Tensioner Mobilisation Technique on Sympathetic Nervous System Function: A Randomised Controlled Trial
Brief Title: Comparative Effects of the Neurodynamic Slider and Tensioner Mobilisation Techniques on Sympathetic Nervous System Function: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Charalambos Papacharalambous, Principal Investigator, European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EEBK/EΠ/2021/58
Record Dates: First submitted 2023-10-11; First posted 2023-10-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Health Care Acceptor
Keywords: Neurodynamic; Neuromobilisation; Tensioner Neurodynamic Technique; Slider Neurodynamic Technique; Slump Test
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sliding Technique Group (Experimental): Participants in the sliding technique group first adopted the SSP. The therapist main-tained the head in a less flexed and closer to neutral position. During this process, they performed full dorsiflexion of the foot, ensuring that the movements allowed the nerve to glide through its pathway rather than creating significant tension
  Interventions: Other: Neurodynamic
- Tension Technique Group (Experimental): Participants in the tensioner technique group first adopted the SSP, then proceeded to enhance neural tension by simultaneously fully dorsiflexing the foot and fully flexing the cervical spine forward, thereby increasing tension throughout the nerve pathway. The technique is applied dynamically with relaxation intervals to prevent any potential negative effects on neural vasculature
  Interventions: Other: Neurodynamic
- Control Group (No Intervention): In this group the participants will be requested to position themselves on the plinth in supine line position. All participants in this group will not receive any intervention and they will be instructed to remain in this position for 20 minutes.

INTERVENTIONS:
Other: Neurodynamic — Neurodynamic Slider and Tensioner Technique
  Arms: Sliding Technique Group; Tension Technique Group

SUMMARY:
In accordance with an independently matched group design methodology, 90 healthy volunteers (aged 18 to 40) were enlisted and randomly assigned to one of three experimental groups (sliding, tension, or control groups). The participants' group assignment was concealed from them. Using the Biopac MP36 electrodermal amplifier, constant skin conductors (SC) levels were captured for 20 minutes. A blind data collector used the Biopac software to gather the data. A pre and post-treatment measurement was taken with the thermal-camera and an ambulatory blood pressure monitor.

DETAILED DESCRIPTION:
Ninety healthy volunteer participants were randomly allocated to three groups (sliding neurodynamic techniques (NDT), tension NDT, and control) using the hypothetico-deductive method of theory testing that allows the comparison within the variables. Additionally, a double-blind experimental research strategy was used in this study. The study's participants were not informed on their allocation to the groups in an effort to reduce the likelihood of expectation bias. It is crucial to note that the researcher maintained his or her blindness throughout the data selection process in order to safeguard the study's internal validity. Two people carried out the experiment in order to accomplish this: the "therapist" who applied the NDT and the "data collector" in charge of documenting the outcomes of the intervention.

Any changes in the Sympathetic Nervous System (SNS) were noted and recorded using three valuable outcome measure tools: the Biopac Galvanic skin response 100B electrodermal activity amplifier (MP36 Biopac Systems Incorporation), a thermo-camera © and an ambulatory blood pressure monitor.

The practical room was set up during the experiment so that neither the therapist nor the subjects came in contact with the apparatus. In order to ensure blinding from the results as the experiment was running, the plinth (treatment area) was separated from the data collection table with the computer and equipment (Biopac, blood pressure monitor, environmental thermometer, and thermo-camera) by a screen. Only the data collector has access to the Biopac software, blood pressure monitor, environmental thermometer, and thermo-camera in order to blind the therapist to the results of the experiment completely. Throughout the whole experiment, the therapist stayed hidden behind the screen.

The therapist begins standardising the equipment when the subjects are seated on the plinth. The thermo-camera has to be positioned correctly, pointing at the participant's hold body in the first stage. Second, the therapist placed the blood pressure monitor's cuff on the participant's left arm. The ideal placement of the skin electrodes was the next step. Each participant's second and third toes on both legs received skin electrodes. When the participant finally assumed their position, the therapist asked the data collector to quickly verify SC activity using the thermo-camera, ambulatory blood pressure monitor, and graph readings from the Biopac acquisition programme.

The experiment comprised three phases: (1) Pre-Intervention Phase, (2) Intervention Phase, and (3) Post-Intervention Phase. The experiment started with an 8-minute stabilisation phase aiming to achieve a physiological resting state, followed by the baseline recording period, which lasted 2 minutes. During this phase, the therapist took the body temperature and the blood pressure of each participant, using the blood pressure monitor and the thermo-camera ©. Following, three phases of 1-minute interventions were applied on the 'intervention leg', each separated by a 1-minute rest period. Finally, the experiment concluded with a 5-minute resting period. The SC was recorded through the Biopac software the whole time, and the whole experiment lasted 20 minutes. Throughout the experiment, the data collector indicated the time frame for each phase with the verbal cue 'Intervention Phase 1 or 2 or 3'.

Moreover, the data collector placed markers on the Biopac graph to demonstrate the start and end of each intervention phase. Finally, when the experiment passed into the Post-Intervention Phase, the therapist took the body temperature and the blood pressure from each participant. It must be noted that NDT manoeuvres during the experiment were performed on the participants as described by Shacklock (2005).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 40 years
2. Body Mass Index less than 30

Exclusion Criteria:

1. Previous History of Lower Back Pain
2. Skin Disorders
3. Previous Experience of Spinal Manual Therapy Treatment
4. Previous Lower Limb Injuries or Trauma
5. Food, Caffeine, Nicotine, or Alcohol consumed 3 hours before the experiment strenuous Activity done 3 hours before the experiment
6. Chronic Systemic Health Conditions (for example, diabetes)
7. Psychiatric Illnesses or Anxiety Disorders
8. Medication that may have an affect on the SNS (for example, anti-depressants, anti-nausea medication, beta-blockers, muscle relaxants)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Biopac Galvanic skin response 100B electrodermal activity amplifier (MP36 Biopac Systems Incorporation) | 7 min continuously monitoring will take place during the intervention (7 min following the start of the experiment).
  The skin electrodes were placed on the 2nd and 3rd toes on both legs of each participant. Aiming to be sure of the maximum contact of the pads sticking on the skin, the ventral surfaces on the 2nd and 3rd toes were initially cleaned with an isopropyl alcohol tissue before the pads were placed. They remained for a few seconds to dry, aiming to remove any sweat residue or unwanted skin that might influence the data reading process.
Thermo-Camera | Monitoring will start when participants will take the final sympathetic slump position on the plinth before the intervention (4 min following the starting of the experiment) and following the intervention (20 min following the start of the experiment).
  Skin temperature will be measured using a thermo-camera (ThermaCam SC2000©, FLIR, Danderyd, Sweden) pre-post intervention. The thermo-camera will be positioned, pointing at the participant's entire body and monitoring the body temperature in degrees Celsius.
Ambulatory blood pressure monitoring | Monitoring will start when participants will take the final sympathetic slump position on the plinth before the intervension (3 min following the starting of the experiment) and following the intevension (18 min following the start of the experiment).
  Therapist placed the cuff of an ambulatory blood pressure monitor (Omron© HEM-9210T Healthcare, Co, Ltd, Kyoto, Japan) on the left arm of the participant. The monitor was used to monitor pre and post-intervention systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- European University Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No